CLINICAL TRIAL: NCT00365235
Title: Genetic Susceptibility to Common Lipid Disorders in Mexico
Brief Title: Understanding the Genetic Basis of Familial Combined Hyperlipidemia in Mexican Individuals
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Paivi Pajukanta, Professor, University of California, Los Angeles
Other Study IDs: 1348; R01HL082762-01A1 (NIH)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Hyperlipidemia, Familial Combined; Coronary Disease
MeSH Terms: conditions — Hyperlipidemia, Familial Combined; Coronary Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood sample is taken from all participants and adipose tissue sample from a subgroup.

SUMMARY:
Familial combined hyperlipidemia (FCHL) is an inherited disorder characterized by elevated levels of cholesterol and triglycerides; it often occurs in Mexican individuals with coronary heart disease (CHD). The purpose of this study is to identify the specific genes that predispose Mexican individuals to FCHL.

DETAILED DESCRIPTION:
CHD is the leading cause of death in Mexico. Dyslipidemia that is characterized by high total cholesterol, high triglycerides, and low "good" high-density lipoprotein (HDL) cholesterol is a risk factor for developing CHD. Research has shown that the Mexican population has an increased tendency towards dyslipidemia, but it is not known what genetic factors contribute to this predisposition. This study will examine the genetic basis of FCHL, which is an inherited form of dyslipidemia characterized by elevated levels of total cholesterol and triglycerides. FCHL is a major contributing factor in CHD; 20% of individuals with CHD under the age of 60 have FCHL. The purpose of this study is to identify and characterize the specific DNA sequence variations that predispose Mexican individuals to FCHL. Results of this study may aid in the development of appropriate prevention and screening techniques.

This study will enroll individuals in Mexico who have FCHL. Participants will attend one study visit for blood collection and DNA sampling. Family members of participants will be contacted and asked to provide a DNA sample also. A select group of participants will return for a second study visit for RNA sampling. Study researchers will analyze participants' DNA and RNA samples, as well as two FCHL genes identified in previous research studies.

ELIGIBILITY:
Inclusion Criteria:

* Elevated levels of serum total cholesterol, triglycerides, or both
* Elevated levels of serum apolipoprotein B (using the Mexican population percentiles)

Exclusion Criteria:

* Tendon xanthomas
* Kidney disease
* Thyroid disorder

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects are Mexicans visiting the Dyslipidemia Clinic at the Instituto Nacional de Ciencias Medicas y Nutricion, Salvador Zubiran, Mexico City, and their family members
Sampling Method: Non-Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2006-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Identifying the specific genes that predispose Mexican individuals to FCHL | Measured through the use of genetic samples

CONTACTS AND LOCATIONS:
Overall Officials: Paivi E. Pajukanta, MD, PhD, Principal Investigator — David Geffen School of Medicine at UCLA, Department of Human Genetics
Locations (1):
- Instituto Nacional De Ciencias Medicas y Nutricion, Mexico City, Mexico